CLINICAL TRIAL: NCT04201340
Title: Topcon DRI OCT Triton With SS-OCT Angio Software Evaluation Study
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Triton OCT-A
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Fluorescein Angiography Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects Presenting with Normal Eyes: Subjects with no known ocular diseases will be imaged on the DRI OCT Triton with SS-OCT Angio software, Zeiss Cirrus HD-OCT 5000, and TRC-50DX
  Interventions: Device: DRI OCT Triton with SS-OCT Angio software; Device: Cirrus HD-OCT 5000; Device: TRC-50DX
- Subjects with retinal pathology present in the vasculature: Subjects with retinal pathology likely to present in the vasculature will be imaged on the DRI OCT Triton with SS-OCT Angio software, Zeiss Cirrus HD-OCT 5000, and TRC-50DX
  Interventions: Device: DRI OCT Triton with SS-OCT Angio software; Device: Cirrus HD-OCT 5000; Device: TRC-50DX

INTERVENTIONS:
Device: DRI OCT Triton with SS-OCT Angio software — The Topcon DRI OCT Triton with SS-OCT Angio software is an OCT with a fundus camera used for diagnostic purposes
Device: Cirrus HD-OCT 5000 — The Zeiss Cirrus HD-OCT 5000 is an OCT used for diagnostic purposes
Device: TRC-50DX — The TRC-50DX retinal camera images the fundus used for diagnostic purposes

SUMMARY:
Comparisons for vascular structure visualization in the retina and choroid.

ELIGIBILITY:
NORMAL GROUP Inclusion Criteria

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects who have not participated in the DRI OCT Triton with SS OCT Angio software Evaluation Prestudy
4. Subjects with normal eye exam bilaterally (laser refractive surgery and cataracts are acceptable)
5. IOP ≤ 21 mmHg bilaterally
6. BCVA 20/40 or better bilaterally

Exclusion Criteria

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT-A scans
3. Subjects with known allergy to fluorescein, or subjects having liver disease, or end-stage renal disease
4. Narrow angle
5. History of leukemia, dementia or multiple sclerosis
6. Concomitant use of hydroxychloroquine or chloroquine
7. Subjects where the study eye was treated after screening and before imaging

RETINAL GROUP Inclusion Criteria

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects who have not participated in the DRI OCT Triton with SS OCT Angio software Evaluation Prestudy
4. BCVA 20/400 or better in the study eye
5. Diagnosis of some type of retinal pathology likely to present in the vasculature in at least one eye as determined by the investigator, may include, but is not limited to: Diabetic retinopathy, Retinal Vein occlusions, Exudative AMD or Macular telangiectasia with expected presentation in the vasculature of, including but not limited to, microaneurysms, capillary dropout and/or choroidal neovascularization.

Exclusion Criteria

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT-A scans
3. Subjects with known allergy to fluorescein or if ICGA is clinically indicated, indocyanine green dyes, shellfish, iodine, or subjects having liver disease, or end-stage renal disease
4. History of leukemia, dementia or multiple sclerosis
5. Concomitant use of hydroxychloroquine or chloroquine
6. Subjects where the study eye was treated after screening and before imaging

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with normal eyes or retinal pathology
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Positive percent agreement (PPA) for each OCT-A device using TRC-50DX as the reference | Day 1
  Comparison of OCT devices to TRC-50DX
Negative percent agreement (NPA) for each OCT-A device using TRC-50DX as the reference | Day 1
  Comparison of OCT devices to TRC-50DX
Agreement of pathology identification between the two OCT-A devices | Day 1
  Compare the pathology identifications between the OCT-A devices

SECONDARY OUTCOMES:
OCT-A image quality score (poor, average and good) | Day 1
  Image quality score

CONTACTS AND LOCATIONS:
Overall Officials: Mayra Tafreshi, Study Director — Topcon Corporation
Locations (1):
- Southeast Retina Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No